CLINICAL TRIAL: NCT03076736
Title: Singing for People With Aphasia (SPA): A Pilot Randomised Controlled Trial of a Group Singing Intervention to Improve Wellbeing
Brief Title: Singing for People With Aphasia
Acronym: SPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1617\014\140293
Record Dates: First submitted 2017-02-28; First posted 2017-03-10 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resource pack (Active Comparator): Aphasia resource pack
  Interventions: Behavioral: Resource pack
- Singing group + resource pack (Experimental): Singing group + Aphasia resource pack
  Interventions: Behavioral: Singing group + resource pack

INTERVENTIONS:
Behavioral: Singing group + resource pack — SPA is a community-based, 10 weekly singing group. Each SPA session comprises 30 minutes of settling in/wrap-up and departure, and 60 minutes of group singing. Sessions will be led by a community music leader, co-facilitated by a person with aphasia, and involve the group singing from a songbook. Musical accompaniment will be provided by the facilitator(s). Small percussion instruments will be available for participants, enabling involvement of those with limited singing ability. Intervention content integrates the Information-Motivation-Behavioural (IMB) skills model of health behaviour change to support individuals in developing the social skills and confidence needed to improve psychosocial outcomes. Participants will also receive the resource pack.
  Arms: Singing group + resource pack
Behavioral: Resource pack — Resource pack with information on living with aphasia and local community activities.
  Arms: Resource pack

SUMMARY:
To undertake a pilot study that will evaluate the feasibility and acceptability of procedures to inform the design and delivery of a definitive RCT of SPA (which would assess the clinical and cost effectiveness of SPA for people with aphasia)

DETAILED DESCRIPTION:
Beyond language function, people with aphasia (PWA) report a range of health problems which negatively affect wellbeing, including reduced confidence and social isolation. These psychosocial outcomes of aphasia are not sufficiently met by healthcare services: improvements in language function do not appear to lead to improvements in wellbeing. National clinical guidelines for stroke reflect this observation and highlight the need for community integration and participation of people with aphasia. This research is about singing groups for people with aphasia (SPA) and is intended to address this need by focusing on the wellbeing and social participation needs of people with aphasia after stroke.

The Investigators engagement activities and early development project provided strong impetus for the proposed study: people with aphasia repeatedly told the investigators that singing in groups may help the participants to reconnect with society, and that this will improve wellbeing.

The investigators have planned a pilot study that will allow an assessment of the extent to which the study processes and the singing groups themselves are feasible to run and are acceptable to participants. The information from this work will help the investigators to decide whether to conduct a larger randomised controlled trial (RCT) which would be a fair test of whether SPA can improve the lives of individuals with post stroke aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of aphasia after stroke
* Willingness to be randomised to either control or SPA (and able to attend the singing venue)
* Conversational English speaker pre-morbidly
* Capacity to consent (assessed by recruiting team using standard tools)

Exclusion Criteria:

* <18 years old
* Currently engaged in a speech or language therapy programme
* Intention to relocate outside the geographical region during the study
* Current participation in another study involving a lifestyle intervention
* Currently attending a singing/music group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
ICEpop CAPability measure for Adults (ICECAP-A) | Measures change from baseline to 3 months post intervention, change from baseline to 6 months post intervention, and change from 3 months to 6 months post intervention
  A 5-item measure of capability for the general adult (18+) population for use in economic evaluation. It focuses on wellbeing and comprises five attributes: Attachment, Stability, Achievement, Enjoyment, Autonomy.
Stroke and Aphasia Quality of Life Scale (SAQOL - 39) | Measures change from baseline to 3 months post intervention, change from baseline to 6 months post intervention, and change from 3 months to 6 months post intervention
  A 39-item health-related quality of life measure with 4 subdomains: physical, psychosocial, communication, and energy.
EQ-5D-5L (health-related quality of life states consisting of five dimensions) | Measures change from baseline to 3 months post intervention, change from baseline to 6 months post intervention, and change from 3 months to 6 months post intervention
  A 5-item measure of health-related quality of life (plus EQ-VAS visual analogue scale), that can be used for cost utility analysis.
modified Reintegration to Normal Living (mRNL) | Measures change from baseline to 3 months post intervention, change from baseline to 6 months post intervention, and change from 3 months to 6 months post intervention
  An 11-item measure that captures social participation (e.g. recreation, movement in the community, and interaction in family or other relationships).

SECONDARY OUTCOMES:
Communication Outcome After STroke (COAST) | Measures change from baseline to 6 months post intervention
  A 20-item measure of communication effectiveness for people with any type of communication problem following stroke
Very Short Version of the Minnesota Aphasia test | Measures change from baseline to 6 months post intervention
  A diagnostic tool to identify aphasia type. Comprised of 4 activities: Identifying names, oral reading words, naming pictures, and written spelling. Audio-recorded to allow for diagnosis of aphasia severity.
Service Receipt Inventory | Measures change from baseline to 6 months post intervention
  Record of types and amount of use of health and social care resources including clinical contacts, formal and informal social care. Completed by Assessor drawing on participant and family accounts.
Care related Quality of Life (CarerQoL-7D)48 | Measures change from baseline to 6 months post intervention
  For completion by carers. A 7-item measures of the impact of providing informal care on carers. Utility tariffs to calculate a weighted sum score of the CarerQol-7D are also available.
Adverse incidents | Measured continuously throughout the intervention (for the intervention group only) and also (for all participants) at 3months and 6months post intervention.
  Adverse events used to gauge the safety of the intervention

OTHER OUTCOMES:
Recruitment | From the start of participant identification through to participant randomisation, over a period of 8 months
  An assessment of the recruitment to the trial
Retention | From Randomisation through study completion, an average of 36 weeks
  An assessment of the retention rates in the trial
Qualitative Interviews | Interviews to be conducted 3 months post-intervention
  15 Qualitative interviews across the intervention and control groups to discuss individuals' experiences of the trial processes and the intervention. Participants will report on the acceptability of trial and intervention activities
Intervention fidelity (intervention group only): Singing group attendance | During the intervention, up to 10 weeks
  A register of attendance at the singing group
Intervention fidelity (intervention group only): Session adherence | During the intervention, up to 10 weeks
  Group facilitators will record which aspects of the intervention manual have been followed during the group session
Intervention fidelity (intervention group only): Observations | During the intervention, up to 10 weeks
  The research team will observe and record the extent to which the group facilitators are following the key elements of the intervention manual and the participants are adhering to facilitator instructions
Intervention fidelity (intervention group only): Video recordings | During the intervention, up to 10 weeks
  The research team will video-record a selection of singing group sessions to assess facilitator and participant adherence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tarrant M, Carter M, Dean SG, Taylor R, Warren FC, Spencer A, Adamson J, Landa P, Code C, Backhouse A, Lamont RA, Calitri R. Singing for people with aphasia (SPA): results of a pilot feasibility randomised controlled trial of a group singing intervention investigating acceptability and feasibility. BMJ Open. 2021 Jan 13;11(1):e040544. doi: 10.1136/bmjopen-2020-040544. PMID 33441355
- [Derived] Tarrant M, Carter M, Dean SG, Taylor RS, Warren FC, Spencer A, Adamson J, Landa P, Code C, Calitri R. Singing for people with aphasia (SPA): a protocol for a pilot randomised controlled trial of a group singing intervention to improve well-being. BMJ Open. 2018 Sep 10;8(9):e025167. doi: 10.1136/bmjopen-2018-025167. PMID 30206095